CLINICAL TRIAL: NCT05049408
Title: Verification of Saliva MMP-1 as a Strong Diagnostic Marker of Oral Cavity Cancer
Brief Title: Verification of Saliva MMP-1 as a Diagnostic Marker of Oral Cavity Cancer
Status: Completed | Type: Observational
Sponsor: S&T Biomed Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: STBM-CT-OSCC-DIA001
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: Mouth Neoplasms; Head and Neck Neoplasms
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group OSCC: Patients with Oral Squamous Cell Carcinoma (OSCC)
  Interventions: Diagnostic Test: MMP-1 Enzyme Linked Immunosorbent assay (ELISA)
- Group OPMD: Patients with oral potentially malignant disorders (OPMD)
  Interventions: Diagnostic Test: MMP-1 Enzyme Linked Immunosorbent assay (ELISA)
- Group HC: Healthy Control
  Interventions: Diagnostic Test: MMP-1 Enzyme Linked Immunosorbent assay (ELISA)

INTERVENTIONS:
Diagnostic Test: MMP-1 Enzyme Linked Immunosorbent assay (ELISA) — The MMP-1 ELISA is to measure salivary MMP-1 levels of participants

SUMMARY:
The study is designed to measure salivary matrix metalloproteinase-1 (MMP-1) using the enzyme-linked immunosorbent assay (ELISA) we developed previously in patients with oral potentially malignant disorders (OPMD), oral squamous cell carcinoma (OSCC), and healthy participants. The purpose of this study is to evaluate the potential of the newly developed salivary MMP-1 ELISA as an adjunctive tool to aid in diagnosis of OSCC.

ELIGIBILITY:
Inclusion Criteria:

* Group OSCC: patients with lesions of OSCC
* Group OPMD: patients with lesions of OPMD
* Group HC: healthy subjects who are not suffering from any oral lesions and having behaviors of smoking, and/or betel nut chewing

Exclusion Criteria:

* Subjects having personal history of other cancers or severe diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Randomly selected samples whose donors meeting the eligibility criteria from tissue bank
Sampling Method: Probability Sample
Enrollment: 1160 (Actual)
Dates: Start 2011-02-17 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2016-12-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity (both range from 0 to 1, the higher the better) of salivary MMP-1 levels as a diagnostic marker for OSCC | 30 days from initial sample obtained for this study

SECONDARY OUTCOMES:
ROC analysis of non-cancer group versus OSCC patients to find the optimal cutoff as the maximum of Youden's index (calculated as sensitivity + specificity - 1 and ranges from 0 to 1, the higher the better) | 30 days from initial sample obtained for this study

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chi-Mei Medical Center, Tainan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chang YT, Chu LJ, Liu YC, Chen CJ, Wu SF, Chen CH, Chang IY, Wang JS, Wu TY, Dash S, Chiang WF, Chiu SF, Gou SB, Chien CY, Chang KP, Yu JS. Verification of Saliva Matrix Metalloproteinase-1 as a Strong Diagnostic Marker of Oral Cavity Cancer. Cancers (Basel). 2020 Aug 13;12(8):2273. doi: 10.3390/cancers12082273. PMID 32823758